CLINICAL TRIAL: NCT02597374
Title: Exploration du système Des Neurones-miroirs Par Enregistrement EEG du Rythme mu Chez l'Enfant Atteint de lésion cérébrale unilatérale Lors d'Action, d'Observation et d'Imagination d'Action du Membre supérieur. " Action-Observation-EEG "
Brief Title: EEG in Children With Unilateral Cerebral Injury During Action and Action Observation(AOE)
Acronym: AOE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CHU-Promoteur 2015-A00985-44
Record Dates: First submitted 2015-10-22; First posted 2015-11-05 (Estimated); Last update posted 2022-07-28 (Actual); Status verified 2022-07

CONDITIONS: Cerebral Palsy; Child
Keywords: Electroencephalography; mu rhythm; Sensorimotor Cortex; Unilateral Cerebral Palsy; Child
MeSH Terms: conditions — Cerebral Palsy | interventions — Electroencephalography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Experimental (Experimental): A 45 mn EEG for all the participants.
  Interventions: Device: EEG

INTERVENTIONS:
Device: EEG — A 45 mn EEG will be performed in each participants during action and action observation of each hand.

SUMMARY:
To study the reactivity of the mu rhythm during action and action-observation by EEG in children with unilateral cerebral injury.

ELIGIBILITY:
Inclusion Criteria:

* unilateral cerebral injury
* hemiplegia

Exclusion Criteria:

* visual or mental or cognitive impairment
* no health insurance

Ages: 6 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Estimated)
Dates: Start 2015-10 (Actual); Primary Completion 2023-10 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Change measures of mu rhythm desynchronization (i.e. alpha band power) before the action execution or action observation and after the action execution or action observation | one day
  The mu rhythm is a spontaneous sensorimotor rhythm made of neurophysiological oscillations with a frequency between 8 herz and 13 herz (alpha band), beside the sensorimotor cortex. The alpha band is recorded on surface electroencephalography (EEG). The power is the square of the amplitude of the spontaneous oscillations.

CONTACTS AND LOCATIONS:
Overall Officials: NGUYEN THE TICH Sylvie, MD-PHD, Principal Investigator — University Hospital, Angers
Locations (1):
- Chu Angers, Angers, France